CLINICAL TRIAL: NCT02657707
Title: Pivotal Study of the MicroVention, Inc. Carotid Artery Stent System Used in Conjunction With the Nanoparasol® Embolic Protection System for the Treatment of Carotid Artery Stenosis in Patients at Elevated Risk for Adverse Events From Carotid Endarterectomy.(CONFIDENCE Trial)
Brief Title: Evaluation of the Roadsaver Stent Used in Conjunction With the Nanoparasol Embolic Protection System for Carotid Artery Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL11003
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Carotid Artery Stenosis
Keywords: stent; stenosis; artery; carotid
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm, open label (Experimental): To evaluate the safety and effectiveness of MicroVention, Inc. Roadsaver™ Carotid Stent System used in conjunction with the Nanoparasol® embolic protection system for the treatment of carotid artery stenosis in patients with elevated risk for adverse events following carotid endarterectomy.
  Interventions: Device: Roadsaver™ Carotid Artery Stent Device; Device: Nanoparasol® Embolic Protection System

INTERVENTIONS:
Device: Roadsaver™ Carotid Artery Stent Device — The Roadsaver™ carotid artery stent system is indicated for use in patients with significant atherosclerotic disease of the carotid arteries.
Device: Nanoparasol® Embolic Protection System — The Nanoparasol® embolic protection system is indicated for use with a guidewire to contain and remove embolic material (thrombus/debris) while performing angioplasty and stenting procedures in carotid arteries.

SUMMARY:
A prospective, multicenter, single-arm, open label clinical study to evaluate the safety and effectiveness of MicroVention, Inc. Roadsaver™ Carotid Stent System used in conjunction with the Nanoparasol® embolic protection system for the treatment of carotid artery stenosis in patients with elevated risk for adverse events following carotid endarterectomy.

DETAILED DESCRIPTION:
Up to 295 patients will be enrolled for this study. All potential patients being considered for the study should have been diagnosed with significant carotid artery stenosis and be considered a high perioperative risk for carotid endarterectomy.

Patients will be evaluated through screening, pre-procedure, index procedure, post-procedure. Follow-up visits will be completed at 30 days, 6 months, and 12, 24, and 36 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between >21 and ≤80 years of age.
2. Patient is willing and capable of complying with all study protocol requirements, including specified follow-up period and can be contacted by telephone.
3. Patient or authorized legal representative is willing to provide written informed consent prior to enrollment in study.
4. Patient should have been diagnosed with carotid artery stenosis and be considered a high operative risk for carotid endarterectomy.
5. Patient is either:

   * Symptomatic with carotid stenosis ≥50% as determined by angiography using NASCET methodology. Symptomatic is defined as amaurosis fugax ipsilateral to the carotid lesion; TIA or non-disabling stroke within 180 days of the procedure within the hemisphere supplied by the target vessel; or
   * Asymptomatic with carotid stenosis ≥80% as determined by angiography using NASCET methodology.
6. Patient has a target lesion located at the carotid bifurcation and/or proximal ICA.
7. Patient has a single de novo or restenotic (post CEA) target lesion or severe tandem lesions close enough that can be covered by a single Roadsaver™ stent.
8. Patients having a vessel with reference diameters between 3.0 mm and 9.0 mm at the target lesion.

High Risk Inclusion Criteria

For inclusion in the study, a patient must qualify in at least one anatomic or co-morbid high-risk condition, as shown below:

Anatomic High Risk Conditions:

1. Patient has a target lesion at or above the second vertebral body (level of jaw) or below the clavicle.
2. Patient has an inability to extend the head due to cervical arthritis or other cervical disorders.
3. Patient is status/post radiation therapy to the neck.
4. Patient has a prior head and neck surgery in the region of the carotid artery.
5. Patient has spinal immobility of the neck.
6. Patient has the presence of tracheostomy stoma.
7. Patient has laryngeal palsy or laryngectomy.
8. Patient has a hostile neck or surgically inaccessible lesion.
9. Patient has severe tandem lesions.

Co-morbid High Risk Conditions:

1. Patient is ≥70 years of age (maximum 80 years) at the time of enrollment.
2. Patient has NYHA Class III or IV congestive heart failure (CHF) with LVEF <35%.
3. Patient has chronic obstructive pulmonary disease (COPD) with FEV <30%.
4. Patient has unstable angina.
5. Patient has had a recent myocardial infarction (≥30 days prior to stenting procedure).
6. Patient has coronary artery disease with two or more vessels with ≥ 70% stenosis.
7. Patient has planned CABG or valve replacement surgery between 31-60 days after the CAS procedure.
8. Patient requires peripheral vascular surgery or abdominal aortic aneurysm repair between 31-60 days following the CAS procedure.
9. Patient has contralateral laryngeal nerve paralysis
10. Patient has restenosis after a previous CEA.
11. Patient has contralateral occlusion in the ICA as the only comorbid high risk condition.

Exclusion Criteria:

1. Patient has life expectancy of less than one year.
2. Patient is experiencing (or has experienced) an evolving, acute, or recent disabling stroke in the last 30 days.
3. Patient has anticipated or potential sources of emboli (e.g. known previously symptomatic patent foramen ovale (PFO), mechanical heart valve, or deep vein thrombosis (DVT) treated within 6 months) that are not adequately treated with antithrombotics for at least two weeks with documented coagulation parameters in the target therapeutic range.
4. Patient has atrial fibrillation.
5. Patient has had an acute myocardial infarction within 60 days prior to index procedure.
6. Patient has had or plans to have any major surgical procedure (i.e. intraabdominal or intrathoracic surgery or any surgery/interventional procedure involving cardiac or vascular system) within 30 days of the index procedure.
7. Patient has a history of major ipsilateral stroke.
8. Patient has >60% carotid stenosis contralateral to the target lesion requiring treatment prior to completion of thes study-required 12 month follow-up.
9. Patient has a modified Rankin Scale of >2 or has another neurological deficit not due to stroke that may confound the neurological patient assessments.
10. Patient has chronic renal insufficiency (serum creatinine ≥2.5 mg/dL) or has a history of severe hepatic impairment, malignant hypertension, and/or is morbidly obese.
11. Patient has platelet count <100,000/μL.
12. Patient has known sensitivity to heparin or previous incidence of Heparin-Induced Thrombocytopenia (HIT) type II.
13. Patient has contraindication to standard of care study medications, including antiplatelet therapy.
14. Patient has known sensitivity to contrast media that cannot be adequately controlled with premedication.
15. Patient has known bleeding diathesis or hypercoagulable state or refuses blood transfusions.
16. Patient has intracranial pathology that, in the opinion of the investigator, makes the patient inappropriate for study participation (e.g. brain tumor, AVM, cerebral aneurysm, cerebral vascular disease [microangiopathy or large vessel], etc.) or would confound neurological evaluation.
17. Patient had intracranial hemorrhage within the last 90 days.
18. Patient is currently enrolled in another investigational study protocol and has not completed its primary endpoint or that will confound the current study endpoints. Patients who are involved in the long-term surveillance of a clinical study are eligible.
19. Patient suffers from confusion or dementia or is unable or unwilling to cooperate with the study requirements and/or follow-up procedures.
20. Patient has a known, unresolved history of drug use or alcohol dependency.
21. Patient has an active infection.
22. Patient has renal failure and/or is on dialysis.
23. Patient has documented uncontrolled diabetes.
24. Patient is pregnant.

Angiographic Exclusion Criteria

A patient is not eligible for enrollment in the study if he/she meets any of the following angiographic exclusion criteria:

1. Patient has a total occlusion of the target carotid arteries (i.e., CCA or ICA).
2. Patient has a previously placed stent in the ipsilateral carotid artery.
3. Patient has severe lesion calcification or vascular tortuosity that may preclude the safe introduction of the sheath, guiding catheter, embolic protection system, or stent.
4. Patient has the presence of mobile filling defect or thrombus in target vessel.
5. Patient has occlusion or presence of "string sign" of the target vessel.
6. Patient has carotid (intracranial) stenosis located distal to target stenosis that is more severe than target stenosis.
7. Patient has known mobile plaque or thrombus in the aortic arch.
8. Patient has a type III aortic arch.
9. Patient in whom femoral access is not possible.
10. Patient has intracranial arteriovenous malformations of the territory of the target carotid artery.
11. Patient has an aneurysm in the territory of the target carotid artery that requires treatment within 12 months.
12. Patient's ipsilateral carotid artery has 2 or more 90 degree bends in the target landing zone.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2016-04-21 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
All stroke, death, and MI | At 30 days
Ipsilateral stroke | At 12 months

SECONDARY OUTCOMES:
Successful deployment of stent | Procedure day
Successful completion of procedure | Procedure day
Successful deployment and retrieval of embolic protection device | Procedure day
Target lesion revascularization (TLR) | At 6 and 12 months
In-stent restenosis | At 6 and 12 months
Major stroke | At 30 days
Minor stroke | At 30 days
Transient ischemic attack (TIA) | Within 30 days
Neurologic death | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Siddiqui, MD, Principal Investigator — University of Buffalo - Neurosurgery; Chris Metzger, MD, Principal Investigator — Wellmont CVA Heart Institute; Peter Schneider, MD, Principal Investigator — Kaiser Permanente Moanalua Medical Center
Locations (37):
- United States (37):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - St. Luke's Medical Center, Phoenix, Arizona
  - Yavapai Regional Medical Center, Prescott, Arizona
  - Kaiser Permanente - Los Angeles, Los Angeles, California
  - San Diego VA Medical Center, San Diego, California
  - Radiology Imaging Associates, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Lyerly Baptist Neurosurgery, Jacksonville, Florida
  - Kaiser Permanente Moanalua Medical Center - Specialty Clinic, Honolulu, Hawaii
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Bryan Heart, Lincoln, Nebraska
  - Darthmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Overlook Medical Center, Summit, New Jersey
  - Albany Medical College, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Feinstein Institute for Medical Research, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - NC Heart and Vascular Research / Rex Hospital, Raleigh, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - University Hospital, Cleveland, Ohio
  - Holy Spirit Cardiology Research, Camp Hill, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Berks Cardiologists, Wyomissing, Pennsylvania
  - Black Hills Cardiovascular Research / Regional Health Hospital, Rapid City, South Dakota
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Methodist Hospital Memphis-Semmes Murphey, Memphis, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor Scott White Health, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Multicare Institute for Research and Innovation, Tacoma, Washington